CLINICAL TRIAL: NCT01938638
Title: An Open-label Phase I Dose-escalation Study to Characterize the Safety, Tolerability, Pharmacokinetics, and Maximum Tolerated Dose of BAY1143572 Given in a Once-daily or an Intermittent Dosing Schedule in Subjects With Advanced Malignancies
Brief Title: Open Label Phase I Dose Escalation Study With BAY1143572 in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16519
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Neoplasms
Keywords: Advanced malignancies; TNBC; DLBCL; Gastric cancer
MeSH Terms: conditions — Neoplasms; Stomach Neoplasms | interventions — atuveciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BAY1143572 [continuous] (Experimental): BAY1143572 will be administered from cycle 1, day 1 (C1D1) onwards once daily continuously
  Interventions: Drug: BAY1143572
- BAY1143572 [on/off] (Experimental): BAY1143572 will be administered from C1D1 in a 3 days on/4 days off schedule
  Interventions: Drug: BAY1143572

INTERVENTIONS:
Drug: BAY1143572

SUMMARY:
The purpose of this study Part A is to determine the safety, tolerability and the pharmacokinetics of BAY1143572 in subjects with advanced malignancies, which are either refractory to or ineligible for treatment with standard agents.

The purpose of this study Part B is:

Determine the safety, tolerability, pharmacokinetics (PK) and maximum tolerated dose (MTDG-CSF) of BAY1143572 with concurrent administration of the granulocyte colony-stimulating factors (G-CSF) in an intermittent and continuous dosing schedule in subjects with advanced malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged >/=21 years
* Dose escalation phase: Subjects with histologically or cytologically confirmed advanced malignancies (solid tumors and malignant lymphomas) who were refractory to or had exhausted all available therapies. Subjects had to have evaluable or measurable disease (as per RECIST 1.1 or Cheson 2007 criteria).
* Expansion phase only: Subjects with advanced, histologically or cytologically confirmed gastric cancer, triple negative breast cancer (TNBC), or diffuse large B-cell lymphoma (DLBCL), who were refractory to or had exhausted all available therapies. Subjects had to have evaluable or measurable disease (as per RECIST 1.1 or Cheson 2007 criteria).
* Archival tumor tissue to conduct molecular and / or genetic studies must be collected from all study subjects enrolled in this study.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Life expectancy of at least 12 weeks
* Adequate bone marrow, liver, and renal functions as assessed by laboratory analysis to be conducted within 7 days prior to the first dose of study drug
* International normalized ratio (INR) and partial thromboplastin time (PTT) </=1.5 times ULN (upper limit of normal)

Exclusion Criteria:

* Known hypersensitivity to the study drug or excipients of the preparation or any agent given in association with this study
* History of cardiac disease including congestive heart failure > New York Heart Association (NYHA) Class II, unstable angina (anginal symptoms at rest) or new-onset angina (within the last 6 months) or myocardial infarction within the past 6 months and cardiac arrhythmias requiring anti-arrhythmic therapy except for beta-blockers and digoxin; evidence for uncontrolled coronary artery disease (e.g. angina pectoris, myocardial infarction within 6 months prior to study entry, major regional wall motion abnormalities upon baseline echocardiography)
* Previous pulmonary embolism within 12 months prior to study entry
* Uncontrolled hypertension defined as systolic blood pressure >150 mmHg or diastolic blood pressure >90 mmHg on 2 or more consecutive blood pressure readings, despite optimal medical management
* Moderate or severe hepatic impairment, i.e. Child-Pugh class B or C
* Known history of human immunodeficiency virus (HIV) infection
* Chronic or active hepatitis B or C, requiring antiviral therapy
* Active clinically serious infections of > Grade 2 and/or active infections that require treatment with systemic agent
* Uncontrolled seizure disorder requiring therapy (such as steroids or anti-epileptics with significant CYP interaction)
* Evidence or history of bleeding disorder, i.e. any hemorrhage / bleeding event of > Grade 2 within 4 weeks prior to the first dose of study drug

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-09-26 (Actual); Primary Completion 2016-08-17 (Actual); Study Completion 2016-09-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Up to 2 years
Maximum tolerated dose (MTD) of BAY1143572 | Up to 1 year
  In Part A: Maximum tolerated dose (MTD) of BAY1143572 In Part B; Maximum tolerated dose ( MTD) with G-CSF of BAY114357 The MTD is defined as the highest dose that can be given such that not more than 20% of subjects experience a dose limiting toxicity (DLT) during cycle 1.

SECONDARY OUTCOMES:
Maximum total drug concentration (Cmax) | Cycle 1, Day 1 and Day 15 (each cycle is 28 days)
Area under the plasma concentration-time curve from time zero to 24 hours (AUC(0-24) | Cycle 1, Day 1 and Day 15 (each cycle is 28 days)
Area under the plasma concentration-time curve from time zero to infinity (AUC) | Cycle 1, Day 1 and Day 15 (each cycle is 28 days)
Time of maximum observed concentration (tmax) | Cycle 1, Day 1 and Day 15 (each cycle is 28 days)
Tumor response based on RECIST 1.1 or Cheson 2007 criteria | Up to 100 weeks
Biomarker evaluation by determination of MYC protein expression and PCNA mRNA | Cycle 1, Day 1, Day 8 and Day 15 (each cycle is 28 days)
  PCNA: proliferating cell nuclear Antigen mRNA: messenger ribonucleic acid

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (9):
- United States (6):
  - Fayetteville, Arkansas
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Hackensack, New Jersey
  - New York, New York
  - Charleston, South Carolina
- Singapore, Singapore
- Seoul, South Korea
- Taipei, Taiwan